CLINICAL TRIAL: NCT03990948
Title: Hepcidin Behavior in Patients With Obesity and Bariatric Surgery
Acronym: HOBS
Status: Terminated | Type: Observational
Why Stopped: Terminated early
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S62085
Record Dates: First submitted 2019-06-17; First posted 2019-06-19 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2022-10

CONDITIONS: Hepcidin
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with obesity: In 100 patients with obesity, blood samples will be collected.
  Interventions: Other: Blood sampling
- Patients with a Sleeve Gastrectomy: In 100 patients with a Sleeve Gastrectomy, blood samples will be collected.
  Interventions: Other: Blood sampling
- Patients with a Roux-en-Y Gastric Bypass: In 100 patients with a Roux-en-Y Gastric Bypass, blood samples will be collected.
  Interventions: Other: Blood sampling

INTERVENTIONS:
Other: Blood sampling — Blood sample collection

SUMMARY:
Iron deficiency is one of the most common nutritional problems observed in patients with obesity and after bariatric surgery. From a therapeutic point of view, iron deficiency can lead to iron deficiency anemia. Iron supplementation carries the risk of exacerbating infections, altering the gut microbiome and iron overload. Therefore, it would be beneficial to use iron supplementation only in truly iron deficient patients. To date, different studies have observed that hepcidin could be a possible indicator of iron status and absorption in different patient populations. Furthermore, it could be used to distinguish anemia due to iron deficiency from inflammation and globin disorder related anemia. How hepcidin concentrations variate in patients with obesity and after bariatric surgery remains unsure.

DETAILED DESCRIPTION:
During the visit in the obesity clinic, eligible patients will be approached for participation by the sub-investigator. Interested patients will receive information regarding the study and receive the information sheet containing the informed consent form. After signing the informed consent form, general information will be collected regarding medical and demographic data using a short questionnaire. Additional questionnaires regarding demographics and menstrual cycle will be collected. Anthropometric measurements will be collected for the determination of the length, weight, hip circumference, waist circumference and body composition. Finally, blood samples will be collected for the determination of iron and inflammation related markers.

ELIGIBILITY:
Inclusion Criteria:

* The patient has to be 18 years or older
* Written informed consent has to be obtained after being informed on all aspects of the study
* The patient has a BMI > 30 kg/m² OR There has to be at least one year between the primary RYGB and the participation in the study OR There has to be at least one year between the primary SG and the participation in the study

Exclusion Criteria:

* Patients younger than 18 years old
* Women who are pregnant or are breastfeeding
* Post-menopausal women, defined as at least 6 months of amenorrhea after the final menstrual period
* Inability to follow the procedures of the studies due to language problems
* Patients who have had more than one bariatric surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with obesity, patients with a Sleeve Gasterctomy or patients with a Roux-en-Y Gastric Bypass
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2019-01-08 (Actual); Primary Completion 2023-12-12 (Actual); Study Completion 2023-12-12 (Actual)

PRIMARY OUTCOMES:
Serum hepcidin concentration | Study visit 1 day
  Serum hepcidin concentration

SECONDARY OUTCOMES:
Hemoglobin concentration | Study visit 1 day
  Hemoglobin concentration
Mean corpuscular volume | Study visit 1 day
  Mean corpuscular volume
Iron concentration | Study visit 1 day
  Iron concentration
Ferritin concentration | Study visit 1 day
  Ferritin concentration
Transferrin concentration | Study visit 1 day
  Transferrin concentration
Transferrin saturation | Study visit 1 day
  Transferrin saturation
C-reactive protein | Study visit 1 day
  C-reactive protein
Vitamin B12 concentration | Study visit 1 day
  Vitamin B12 concentration
Folate (RBC level) | Study visit 1 day
  Folate (RBC level)
Folate (serum level) | Study visit 1 day
  Folate (serum level)

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided